CLINICAL TRIAL: NCT01041729
Title: Phase IV Study of Statins for Assess the Long-term Pleiotropic Effect Upon Nitric Oxide and C-Reactive Protein Levels in Patients With Peripheral Arterial Disease
Brief Title: Long-term Pleiotropic Effect of Statins in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Joaquin de Haro, M.D., Hospital Universitario Getafe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STA-2009 NO-CRP
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): Patients with Peripheral Arterial Disease in Fontaine Stage II treated with Atorvastatin 40mg/day during 12 months
  Interventions: Drug: Atorvastatin
- Control (Active Comparator): Patients with Peripheral Arterial Disease in Fontaine Stage II without treatment with Atorvastatin 40mg/day during 12 months.
  Standard Medical Treatment
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Drug: Atorvastatin — Patients with Peripheral Arterial Disease in Fontaine Stage II treated with Atorvastatin 40mg/day during 12 months
  Arms: Atorvastatin
Drug: Standard Medical Treatment — Patients with Peripheral Arterial Disease in Fontaine Stage II without treatment with Atorvastatin 40mg/day during 12 months.
  Standard Medical Treatment.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the long-term effects of statins, atorvastatin, upon Nitric Oxide, as an endothelial function assessment, and C-Reactive Protein, an inflammatory marker, levels in patients with Peripheral Arterial Disease. These long-term biological pleiotropic effects of statins will offer information on the role of endothelial function and systemic inflammation in the etiopathogenesis of PAD.

ELIGIBILITY:
Inclusion Criteria:

* patients at the time of diagnosis of Fontaine grade II peripheral arterial disease (PAD), confirmed by hemodynamic evaluation (Doppler ultrasound)
* over 18 years old

Exclusion Criteria:

* patients had previously undergone revascularization
* patients were receiving treatment with statins
* patients with contraindications to statin use.
* patients with coexistence of chronic inflammatory diseases or steroidal medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
High-sensitivity C-Reactive Protein (hsCRP) and nitrites plasma levels at baseline and after one month and one year of inclusion. | Baseline and after one month and one year of inclusion.

SECONDARY OUTCOMES:
Lipid profile | baseline and after one month and one year of inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin De Haro, M.D., Principal Investigator — Hospital Universitario Getafe
Locations (1):
- Hospital Universitario Getafe, Getafe, Madrid, Spain